CLINICAL TRIAL: NCT06617208
Title: Prognostic IntraOperative Biomarkers ideNtification in Tumor rElatEd suRgery (PIONEER Study)
Brief Title: Prognostic IntraOperative Biomarkers ideNtification in Tumor rElatEd suRgery
Acronym: PIONEER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Koen van der Kuil, PhD Student, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PaNaMa 12744
Record Dates: First submitted 2024-09-12; First posted 2024-09-27 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Glioma; Glioblastoma (GBM); Brain Tumor-Glioma
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neuropixel probe recording (Experimental): Cortical electrophysiology using the Neuropixel probe is performed to record brain activity in the peritumoral cortex
  Interventions: Device: Neuropixel probe recording

INTERVENTIONS:
Device: Neuropixel probe recording — Neuropixel recordings captures neuronal activity at the single-neuron level across the layers of the cortex.
  Other Names: laminar electrophysiology; cortical depth electrophysiology

SUMMARY:
INTRODUCTION AND RATIONALE

Aggressive brain tumors like glioma have the ability to infiltrate the surrounding healthy brain tissue, disrupting normal neuronal activities and leading to impaired motor and cognitive functions, as well as causing epilepsy. This malignant brain tumor is considered one of the most challenging cancers to treat, with a median survival of 12 to 15 months. Recent findings on direct neuron-tumor interactions indicate that abnormal brain activity in the regions surrounding brain tumors may contribute to develop epilepsy and accelerating tumor growth. Tumors tend to 'fuel' themselves with neurotransmitters released during its 'daily' neuronal firing. Hyperactive neurons in the peritumoral cortex can form excitatory electrochemical synapses with surrounding tumor cells, creating direct communication pathways within the peritumoral microenvironment, which aids in the progression and proliferation of tumor cells via direct and paracrine signalling pathways. However, the specific features of this abnormal brain activity in the peritumoral cortex have not been fully clarified and information on the pathological changes of neuronal activity in glioma patients is largely lacking. To advance more effective treatment strategies, it is crucial to better understand the complex interactions between the tumor and the brain.

This is especially important for the group of patients of which many perceive diminished quality of life because of epilepsy, cognitive functioning and language problems after tumor surgery. Furthermore, a thorough understanding is lacking of what tumor resection does to the original hyperactive peritumoral cortex and if resecting this is beneficial for improving postoperative outcome both for epilepsy as well as regarding survival. Therefore, identifying the hyperactive peritumoral cortex and directly addressing its impacts on the brain function and long-term surgical outcome could be a promising novel therapeutic strategy for treating glioma patients.

STUDY AIM

The measurement focuses on capturing neuronal activity at single-neuron resolution in the peritumoral cortex of glioma patients using cortical depth electrodes. It is well-established that gliomas can remodel the surrounding brain tissue, leading to abnormal neuronal hyperactivity, which contributes to tumor progression and epilepsy. However, the specific neuronal patterns and underlying mechanisms of these changes are not yet fully understood. This study will aim to collect detailed single-neuron recordings in this context, enabling us to map the precise neurophysiological disruptions caused by gliomas. On the long term, this research could lay the groundwork in identifying novel therapeutic approaches by providing critical in-sights into how gliomas alter brain function.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 yrs and 90 yrs old with radiologically diagnosed GBM
* Eligible for surgery according to standard practices. If suitable and necessary according to standard practices, awake surgery is also permitted.
* Written Informed consent.

Exclusion Criteria:

* Inability to give consent because of or language barrier
* Psychiatric history
* Previous brain tumour surgery or radiotherapy
* Severe aphasia or dysphasia
* Patient has pacemaker or other implanted electrical device such as vagal nerve stimulator or other

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of Successful Neuropixels Probe Recordings During Glioma Surgeries | From the beginning to end of tumor surgery
  Description:
  The primary outcome measure is the number of successful Neuropixels depth electrode recordings achieved during glioma surgeries. Success is defined as:
  Sterility: No postoperative infections, assessed by clinical follow-up and microbiological testing.
  Signal Quality: Signal-to-noise ratio (SNR) above 30 dB, as measured during and after surgery through electrophysiological software.
  Device Integrity: No fractures or damage to the Neuropixels probe, verified by post-procedure inspection.
  Training Efficiency: Setup time and error reduction during the recording process, recorded across surgeries to assess team proficiency.

SECONDARY OUTCOMES:
Prognostic Biomarker Identification (Unit: Number of Isolated Single Neurons with Tumor-Modulated Activity): | From the beginning to end of surgery
  The secondary outcome will focus on identifying prognostic biomarkers through intra-operative recordings using Neuropixels. This includes measuring the number of single neurons isolated with distinct spiking or waveform characteristics that correlate with tumor pathology. The outcome will be quantified as the number of neurons showing unique tumor-related activity patterns (e.g., altered firing rates, waveform morphology) across patients undergoing surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Eelkman Rooda, MD PhD, Study Director — Erasmus Medical Center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Coughlin B, Munoz W, Kfir Y, Young MJ, Meszena D, Jamali M, Caprara I, Hardstone R, Khanna A, Mustroph ML, Trautmann EM, Windolf C, Varol E, Soper DJ, Stavisky SD, Welkenhuysen M, Dutta B, Shenoy KV, Hochberg LR, Mark Richardson R, Williams ZM, Cash SS, Paulk AC. Modified Neuropixels probes for recording human neurophysiology in the operating room. Nat Protoc. 2023 Oct;18(10):2927-2953. doi: 10.1038/s41596-023-00871-2. Epub 2023 Sep 11. PMID 37697108
- [Background] Paulk AC, Kfir Y, Khanna AR, Mustroph ML, Trautmann EM, Soper DJ, Stavisky SD, Welkenhuysen M, Dutta B, Shenoy KV, Hochberg LR, Richardson RM, Williams ZM, Cash SS. Large-scale neural recordings with single neuron resolution using Neuropixels probes in human cortex. Nat Neurosci. 2022 Feb;25(2):252-263. doi: 10.1038/s41593-021-00997-0. Epub 2022 Jan 31. PMID 35102333
- [Background] Chung JE, Sellers KK, Leonard MK, Gwilliams L, Xu D, Dougherty ME, Kharazia V, Metzger SL, Welkenhuysen M, Dutta B, Chang EF. High-density single-unit human cortical recordings using the Neuropixels probe. Neuron. 2022 Aug 3;110(15):2409-2421.e3. doi: 10.1016/j.neuron.2022.05.007. Epub 2022 Jun 8. PMID 35679860
- [Background] Leonard MK, Gwilliams L, Sellers KK, Chung JE, Xu D, Mischler G, Mesgarani N, Welkenhuysen M, Dutta B, Chang EF. Large-scale single-neuron speech sound encoding across the depth of human cortex. Nature. 2024 Feb;626(7999):593-602. doi: 10.1038/s41586-023-06839-2. Epub 2023 Dec 13. PMID 38093008
- [Background] Krishna S, Choudhury A, Keough MB, Seo K, Ni L, Kakaizada S, Lee A, Aabedi A, Popova G, Lipkin B, Cao C, Nava Gonzales C, Sudharshan R, Egladyous A, Almeida N, Zhang Y, Molinaro AM, Venkatesh HS, Daniel AGS, Shamardani K, Hyer J, Chang EF, Findlay A, Phillips JJ, Nagarajan S, Raleigh DR, Brang D, Monje M, Hervey-Jumper SL. Glioblastoma remodelling of human neural circuits decreases survival. Nature. 2023 May;617(7961):599-607. doi: 10.1038/s41586-023-06036-1. Epub 2023 May 3. PMID 37138086
- [Background] Venkataramani V, Yang Y, Schubert MC, Reyhan E, Tetzlaff SK, Wissmann N, Botz M, Soyka SJ, Beretta CA, Pramatarov RL, Fankhauser L, Garofano L, Freudenberg A, Wagner J, Tanev DI, Ratliff M, Xie R, Kessler T, Hoffmann DC, Hai L, Dorflinger Y, Hoppe S, Yabo YA, Golebiewska A, Niclou SP, Sahm F, Lasorella A, Slowik M, Doring L, Iavarone A, Wick W, Kuner T, Winkler F. Glioblastoma hijacks neuronal mechanisms for brain invasion. Cell. 2022 Aug 4;185(16):2899-2917.e31. doi: 10.1016/j.cell.2022.06.054. Epub 2022 Jul 31. PMID 35914528
- [Background] Venkataramani V, Tanev DI, Strahle C, Studier-Fischer A, Fankhauser L, Kessler T, Korber C, Kardorff M, Ratliff M, Xie R, Horstmann H, Messer M, Paik SP, Knabbe J, Sahm F, Kurz FT, Acikgoz AA, Herrmannsdorfer F, Agarwal A, Bergles DE, Chalmers A, Miletic H, Turcan S, Mawrin C, Hanggi D, Liu HK, Wick W, Winkler F, Kuner T. Glutamatergic synaptic input to glioma cells drives brain tumour progression. Nature. 2019 Sep;573(7775):532-538. doi: 10.1038/s41586-019-1564-x. Epub 2019 Sep 18. PMID 31534219